CLINICAL TRIAL: NCT06735430
Title: Ciprofol Based on Total Intravenous Anesthesia During Pediatric Laparoscopic Surgery: a Prospective, Double-blind, Randomized Controlled, Non Inferiority Clinical Trial
Brief Title: Ciprofol Based on Total Intravenous Anesthesia During Pediatric Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, Doctor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Tongji Hospital-20241204
Record Dates: First submitted 2024-12-04; First posted 2024-12-16 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Hernia; Laparoscopic Surgery; Appendicitis, Surgery
Keywords: Ciprofol; Propofol; Total Intravenous Anesthesia; Children
MeSH Terms: conditions — Appendicitis | interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ciprofol (Experimental): Ciprofol for anesthesia induction (0.5mg / kg) and anesthesia maintenance (1-2.5mg/ (kg·h))
  Interventions: Drug: Ciprofol
- Propofol (Other): Propofol for anesthesia induction (2mg / kg) and maintenance of anesthesia (4-10 mg / (kg·h))
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ciprofol — Ciprofol for anesthesia induction (0.5mg / kg) and anesthesia maintenance (1-2.5mg/ (kg·h))
  Arms: Ciprofol
Drug: Propofol — Propofol for anesthesia induction (2mg / kg) and maintenance of anesthesia (4-10 mg / (kg·h))
  Arms: Propofol

SUMMARY:
a prospective, double-blind, fully randomized controlled, non-inferiority clinical trial to investigate the use of total intravenous anesthesia in pediatric laparoscopic surgery.

DETAILED DESCRIPTION:
Ciprofol is a better alternative to surgical sedatives. The clinical application basis of Ciprofol in pediatric anesthesia is still lacking. Therefore, the investigators designed a prospective, double-blind, fully randomized controlled, non-inferiority clinical trial to investigate the use of all-through intravenous anesthesia in pediatric laparoscopic surgery. Our main hypothesis is that in pediatric surgery, using Ciprofol by intravenous anesthesia, the extubation time is no longer than that the propofol group.

ELIGIBILITY:
Inclusion Criteria:

* laparoscopic surgery under general anesthesia

Exclusion Criteria:

* Known allergies to propofol and ciprofol,
* Mental retardation, cognitive and affective disorders, psychiatric or neurological disorders;
* uncooperate with peripheral venipuncture and catheterization;
* History of acute upper respiratory tract infection in the past 2 weeks;
* With severe respiratory, circulation, liver and kidney insufficiency;
* Body mass index (BMI) of 30 kg/m² or 15 kg/m²;
* Known long-term use of sedative drugs;
* ASAⅢ grade or above;
* recent participation in other clinical studies.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2025-03-09 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Extubation time | up to 1 hour
  Time interval between drug withdrawal and removal of the tracheal catheter

SECONDARY OUTCOMES:
Aldrete Score | up to 2 hours
  In the PACU, Investigators using Aldrete score scale(0- 10 points)
Emergence Agitation | up to 2 hours
  In the PACU, Investigators assessed emergence delirium using PAED 0-20 points)
Postoperative Pain | 24 hours
  use the FLACC pain score(0- 10 points)
Postoperative nausea and vomiting | 24 hours
  Investigators assessed postoperative nausea and vomiting BARF scale(0-10points)
satisfaction degree | 24 hours
  Child and/or Parent Satisfaction Survey (0-10 points)

CONTACTS AND LOCATIONS:
Overall Officials: mujun Chang, Dr., Study Director — Tongji Hospital
Locations (1):
- Tongji hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No